CLINICAL TRIAL: NCT03839381
Title: Turkish Version of Mini-BESTest- Balance Evaluation Systems Test: A Translation and Transcultural Adaptation Study Incorporating Validity and Reliability Analysis for Adult Participants With Sensoriomotor Impairments
Brief Title: Turkish Version of Mini-BESTest, Validity and Reliability for Adult Participants With Sensoriomotor Impairments
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sema BÜĞÜŞAN ORUÇ, PHD student, Ordu University
Other Study IDs: ORDU345
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease; Multiple Sclerosis; Trauma, Brain
Keywords: mini BESTest; balance defisit; postural control; Sensoriomotor impairment
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to present the Turkish version of miniBESTest which evaluates the reasons of balance deficit and postural control. Accordingly, a practice of validity and reliability on adult patients with sensoriomotor impairments will be performed by utilizing the Turkish version of miniBESTest in this study.

DETAILED DESCRIPTION:
Physical therapists encounter postural control problems frequently. These problems require multifaceted assessment. Therefore, the treatment of postural control problems should be planned after a multifaceted assessment.

Balance Evaluation Systems Test (BESTest) comprises 27 items and evaluate all components of postural control. MiniBESTest is a shortened version of BESTest with 14 tasks. MiniBESTest still addresses almost all components of postural control and can be performed 15 min. MiniBESTest is one of the most common methods which practiced on adult patients.

The aim of this study is to present the Turkish version of miniBESTest which evaluates the reasons of balance deficit and postural control. Accordingly, a practice of validity and reliability on adult participants with sensoriomotor impairments will be performed by utilizing the Turkish version of miniBESTest in this study.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of sensoriomotor impairment Able to walk with or without an assistive device (e.g. walker, cane, ankle-foot orthosis...) Ability to tolerate the balance tasks without fatigue.

Exclusion Criteria:

Severe cognitive or communication impairments Hemodynamic or clinical instability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was planned participants who have sensoriomotor impairments were referred to the Ordu University Educational Research Hospital neurology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-04 (Estimated); Primary Completion 2019-11-29 (Estimated); Study Completion 2019-12-04 (Estimated)

PRIMARY OUTCOMES:
Mini BESTest | 10-15 minutes.
  Mini-BESTest focuses on dynamic balance. It includes a total of 14 different tasks, each rated on a 3-level between 0 (severe postural control impairment) and 2 (no postural control impairment) with a maximal score of 28.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Lemay JF, Roy A, Nadeau S, Gagnon DH. French version of the Mini BESTest: A translation and transcultural adaptation study incorporating a reliability analysis for individuals with sensorimotor impairments undergoing functional rehabilitation. Ann Phys Rehabil Med. 2019 May;62(3):149-154. doi: 10.1016/j.rehab.2018.12.001. Epub 2018 Dec 27. PMID 30594663
- [Background] Horak FB, Wrisley DM, Frank J. The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther. 2009 May;89(5):484-98. doi: 10.2522/ptj.20080071. Epub 2009 Mar 27. PMID 19329772